



**Drug Use Investigation** 

**Protocol** 

Pfizer Japan Inc.

Date prepared: April 8, 2013 (Version 2)

Protocol ID: A0081261

### Introduction

Pregabalin, an active ingredient of Lyrica Capsule (hereinafter called "the product"), is one of the derivatives of γ-aminobutyric acid (GABA) developed at Northwestern University, USA.

In the excessively stimulated excitable nervous system, pregabalin binds with high affinity to  $\alpha 2\delta$  protein (an auxiliary subunit of voltage-gated calcium channels), which supposedly reduces calcium inflow into presynaptic nerve terminals and suppresses the synaptic release of excitatory neurotransmitters, consequently leading to manifestation of analgesic activity.

As of February 2012, the product has been approved for indications of neuropathic pain (peripheral neuropathic pain and central neuropathic pain) and the like in 120 countries of the world, including the US, European Union countries, Australia and Canada. In Japan, the product has been approved for indications of peripheral neuropathic pain in October 2010, pain associated with fibromyalgia in June 2012, and neuropathic pain in February 2013.

The drug use investigation on Lyrica Capsule (hereinafter called "the survey") will be undertaken to collect or check information about the incidence of each type of disorder arising from adverse reactions to the product and the information on quality, efficacy and safety of the product in routine clinical use. The information collected through the survey will be supplied as the information on proper use of the product to medical facilities and used to prepare the application materials for reexamination of the product. To this end, the survey needs to be carried out in compliance with the Good Post-marketing Surveillance Practice (Ministry of Health, Labour and Welfare [MHLW] Ordinance No. 171, dated December 20, 2004). The case data collected through this survey will be reported to the MHLW pursuant to the Pharmaceutical and Medical Device Act. If applicable, the data including names of drugs, adverse reactions, gender and age by decade may be disclosed as a listing of patients in the "Pharmaceuticals and Medical Devices Safety Information" and "Pharmaceuticals and Medical Devices Information Website (http://www.info.pmda.go.jp)" which are issued and managed, respectively, by the MHLW. The collected case data may be also disclosed if the MHLW is requested to disclose them pursuant to the "Act on Access to Information Held by Administrative Organs" (Act No. 42, dated May 14, 1999). In any of the above cases, the report does not cover the name of the physicians, facilities or the like involved, and these pieces of information will never be published or disclosed.



## **Objectives**

The objective of this survey is to evaluate the safety and efficacy of the product in routine clinical practice. In addition, efforts will be made to collect information on the incidence of previously known and unknown adverse reactions that will occur under actual use conditions during the survey period. At the same time, the necessity of conducting a special investigation or a post-marketing clinical study will be evaluated.

The following events will be evaluated as major investigation items;

- Peripheral edema and edema-related events\*
- Dizziness, somnolence, loss of consciousness, syncope and potential for accidental injury
- Vision-related events
- \*: Adverse events of the cardiovascular and respiratory systems will be also checked.

## Study population

The survey covers the patients satisfying all of the following requirements:

- Patients not participating in any other survey or study of the product
- Patients having never used the product before the survey

The indications, dosage and administration of the product are specified below:

Indications: Neuropathic pain\*, pain associated with fibromyalgia\*\*

[Neuropathic pain]

Dosage and Administration: The usual starting dose in adults is 150 mg/day of pregabalin orally administered in 2 divided doses, which may be gradually increased to 300 mg/day over one week or longer. The dose may be adjusted depending on age and symptoms as appropriate. provided the daily dose may not exceed 600 mg and the product should be orally administered in 2 divided doses regardless of the daily dose.

> The latest version of the package insert should be referred to when the product is prescribed.

The survey does not cover pain associated with fibromyalgia.

## Target sample size

The target sample size is 3400 patients with neuropathic pain in total, including 3000 patients with peripheral neuropathic pain (1000 patients with post herpetic neuralgia, if possible, and 2000 patients with peripheral neuropathic pain of the types other than post herpetic neuralgia), and 400 patients with central neuropathic pain (300 patients with post-stroke pain, if possible, and other patients with pain following traumatic spinal cord injury and pain due to Parkinson's disease). For peripheral neuropathic pain, approximately 100 each of patients should be accumulated, if possible, for trigeminal neuralgia, peripheral entrapment neuropathy, jatrogenic neuropathy, neuropathy due to tumor-induced nerve compression or infiltration, posttraumatic pain, and chronic cauda equina syndrome.

[Rationale]



Neuropathic pain to be enrolled in April 2013 and thereafter will cover peripheral neuropathic pain including trigeminal neuralgia, peripheral entrapment neuropathy, iatrogenic neuropathy, neuropathy due to tumor-induced nerve compression or infiltration, posttraumatic pain, and chronic cauda equina syndrome, as well as central neuropathic

The target sample size of 3400 patients with neuropathic pain is expected to have a 97% probability to detect adverse reactions occurring at the incidence of 0.1% or higher in at least 1 patient. Of the adverse reactions included in the major investigation items, vision-related events are anticipated to develop at the lowest incidence during the survey. In clinical studies of the product conducted in Japan and overseas, the lower bound of the 95% confidence interval for the incidence of this adverse reaction was 6.70% (incidence 7.40%, 380/5134 patients). If this adverse reaction develops at the same incidence as in these clinical studies, this reaction is expected to occur in 227 or more of 3400 patients. Since the safety and efficacy of the product should be evaluated in patients with each type of neuropathic pain, enrollment of the following number of patients will be ensured; approximately 100 patients each, if possible, for trigeminal neuralgia, peripheral entrapment neuropathy, iatrogenic neuropathy, neuropathy due to tumor-induced nerve compression or infiltration, posttraumatic pain, and chronic cauda equina syndrome, approximately 300 patients for post-stroke pain, and a certain number of patients for pain following traumatic spinal cord injury and pain due to Parkinson's disease.

This sample size will also allow for adequate evaluation of the characteristics of other adverse reactions included in the major investigation items. The characteristics to be evaluated include time of onset and duration of adverse reactions, and these were also investigated in the clinical studies.

## 4 Planned survey period

The survey period and the period for registration into the survey are specified below:

Survey period\* : January 2011 to April 2017 Registration period : January 2011 to January 2017

\* A contract will be concluded on or after the first day of the survey period, and registration of patients will be subsequently started. Observation of all registered patients will be completed by the last day of the contract period.

## 5 Survey procedures

### 5.1 Survey method

The survey will be conducted with the central registration system. Patient registration will be continued until the number of registered patients reaches the target number.

## 5.2 Data collection method

During this survey, an Internet-based electronic data collection system for post-marketing surveillance will be used for patient registration, survey data entry and data confirmation. PostMaNet of Fujitsu FIP Corporation (hereinafter called "the system") will be utilized for this survey. Security during data transmission will be ensured by authenticating each investigator with individual user ID and password and using the latest protocol for SSL enciphered communication. Detailed procedure and methods for data entry, correction and confirmation are separately specified in the data entry sample etc.

## 5.3 Patient registration

After the user ID and password are issued to each investigator, the investigator will enter the following basic information on the patient registration screen: name initials of the patient (as needed), ID code, gender, birth date, starting date for treatment with the product and eligibility to the survey. Considering that the incidence of adverse events (peripheral edema, dizziness, etc.) was highest during the early stage of treatment with the product in phase 3 studies conducted in Japan, registration of patients should be done within 7 days after the start of treatment with the product, as a rule (within 14 days at latest) to enable appropriate collection of information on these adverse events.



## 5.4 Observation period

The observation period will start on the first day of treatment with the product (Day 1) and last until Week 13 (Day 91). However, in cases where treatment has been completed or discontinued before Week 13, observation will be continued until completion (discontinuation) of treatment, and follow-up will be made for one week (7 days) after completion (discontinuation) of treatment. During this survey, safety will be evaluated on the day of the first visit after the end of the observation period (including the last day of the observation period), as a rule. In cases where treatment has been completed or discontinued, safety will be evaluated until the day of the first visit following 7-day period after the completion (discontinuation) of treatment, and safety information will be collected for this period.



Supplementary note: Completion of treatment means cases where further treatment with the product is judged unnecessary because of achievement of the purpose of treatment set at the start of treatment (e.g., cure of target diseases).

### 5.5 Precautions in data entry, correction and confirmation

### (1) Data entry

The investigator should check each survey item and enter and transmit the data into the system, on the basis of the records of healthcare (medical records, test reports, etc.). Data entry sample etc. should be referred to for detailed procedure.

#### (2) Data correction

If Pfizer Japan Inc. (hereinafter called "the sponsor") places inquiry about the entered information, the investigator should check the above-mentioned healthcare records again and, as needed, correct the once entered data and transmit the corrected data. Data entry sample etc. should be referred to for detailed procedure.

## (3) Data confirmation

Upon completion of entry and correction of all survey data, the investigator should check the survey form and attach his/her electronic signature to it. Data entry sample etc. should be referred to for detailed procedure.

## 6 Items and schedule of survey

The investigator will conduct the survey in accordance with the observation schedule given below. After conclusion of the contract on the survey, the investigator will register eligible patients. Then, the investigator will check the data on each registered patient (including the data on background variables at the start of treatment) and fill in the survey form for each patient.



## Observation schedule

| | | Registration form | Survey form | | | |
|---|---|---|---|---|---|---|
| Time | | - | | Observation period | | |
| Survey ite | ems | At registration | Start of treatment | Week<br>4 | Week 13 | 7 days after completion/ discontinuation*4 |
| | ID code | • | 0 | | | |
| Identifiable | Name initials (not indispensable) | • | 0 | | | |
| patient | Gender | • | 0 | | | |
| information | Birth date | • | 0 | | | |
| | Eligibility | • | 0 | | | |
| | First day of treatment with the product | • | 0 | | | |
| | Target Disease | • | • | | | |
| | Height/body weight *2 | | • | | | |
| | Hospitalization status | | | | | |
| | (inpatient/outpatient) | | | | | |
| | Presence/absence of hepatic/renal | | | | | |
| Background | dysfunction | | | | | |
| variables | Creatinine clearance | | • | | | |
| variables | With or without hemodialysis | | • | | | |
| | Presence/absence of ocular disease | | | | | |
| | history/complications | | | | | |
| | Disease history | | • | | | |
| | History of previous treatment drugs for | | | | | |
| | the target disease *3 | | | | | |
| | Pregnancy status (females only) | | • | | | |
| | eatment with the product | | <b>←</b> | | <b>—</b> | |
| | therapy (drug therapy/non-drug therapy) | | <b>←</b> | | <b></b> | |
| | l findings/laboratory test) | | - | _ | <b>—</b> | |
| (1) Body wei | ght 1. [Presence/absence of peripheral | | • | • | • | |
| (4) Laborator | edema or edema in general], [Presence/absence of dizziness, somnolence, loss of consciousness, syncope or potential for accidental injury], [Presence/absence of ophthalmological abnormalities], [Presence/absence of suicidal ideation (including suicide attempt and suicide after start of treatment)], [Presence/absence of pathologic changes in appetite and activity] 2. [Presence/absence of withdrawal symptom/rebound phenomenon] e/absence of hyperalgesia ry test [(1) Patient-rated pain score | | • | • | • | • |
| Clinical evaluation | (2) Patient-rated sleep disorder score | | • | • | • | |
| | <ul><li>(3) Patient's impression (PGIC)</li><li>(4) Physician's impression (CGIC)</li></ul> | | | | • | |
| Patient summary | | | | | • | |
| Efficacy evaluation | | | | | • | |
| | Adverse events | | <b>—</b> | | <b>—</b> | |

- lacktriangle Data to be entered;  $\bigcirc$  Data to be reflected
- 1) Entry at the time of patient registration. These pieces of information related to patient registration will be transmitted within 7 days after the start of treatment, as a rule, and within 14 days at the latest.
- 2) Body weight at the start of treatment will be entered in the field of "Body weight" in Tests (clinical findings/laboratory test).
- 3) The drugs previously used for the treatment of the target disease during the period from 14 days to 1 day before the start of treatment with the product will be entered.
- 4) In cases where treatment has been completed (discontinued) before the end of the observation period, follow-up is made for one week (7 days) after completion (discontinuation) of treatment.

### 6.1 Background variables

(1) The information at the start of treatment will be entered in the patient registration form.

[1] ID code



- [2] Name initials (as needed)
- [3] Gender
- [4] Birth date
- [5] First day of treatment with the product
- [6] Eligibility
- [7] Target disease

The relevant disease will be selected from the diseases listed below.

Post herpetic neuralgia, painful diabetic neuropathy, other types of peripheral neuropathic pain, various types of central neuropathic pain, others

Table Common disorders included in neuropathic pain [Classification by the site of nerve injury]

(Source: Reference 1)

| Neuropathic pain | |
|---|---|
| Peripheral neuropathic pain | Central neuropathic pain |
| Post herpetic neuralgia | Post-stroke pain |
| Painful diabetic neuropathy | Pain following traumatic spinal cord injury |
| Complex regional pain syndrome | Pain due to multiple sclerosis |
| Chemotherapy-induced neuropathy | Compressive myelopathy due to spinal canal |
| HIV-induced sensory neuropathy | stenosis |
| Phantom pain* | Pain due to Parkinson's disease |
| Trigeminal neuralgia | HIV-induced myelopathy |
| <ul> <li>Acute/chronic inflammatory demyelinating</li> </ul> | Post-ischemic myelopathy |
| polyradiculoneuropathy | Post-radiation myelopathy/post-radiation |
| Alcoholic neuropathy | encephalopathy |
| Peripheral entrapment neuropathy (carpal tunnel) | Syringomyelia/syringobulbia |
| syndrome etc.) | |
| latrogenic neuropathy | |
| (post-mastectomy pain, post-thoracotomy pain, etc.) | |
| Idiopathic sensory neuropathy | |
| Neuropathy due to tumor-induced nerve compression | |
| or infiltration | |
| Neuropathy due to malnutrition | |
| Post-radiation plexopathy | |
| Radiculopathy | |
| Poisoning neuropathy | |
| Post-traumatic pain | |
| Traumatic avulsion injury of the brachial plexus | |
| Glossopharyngeal neuralgia | |
| Autoimmune neuropathy | |
| Chronic cauda equina syndrome | |

May be viewed as both peripheral neuropathic pain and central neuropathic pain.

- (2) The following information at the start of treatment will be entered in the survey form.
  - [1] Height
  - [2] Body weight (information at the start of treatment will be entered in (1) "Body weight" in Section 6.4 Tests.)
  - [3] Hospitalization status (inpatient/outpatient)
  - [4] Target disease (name of the disease or diagnosis requiring use of the product), major site affected, duration of sickness, underlying disease and its duration
  - [5] Presence/absence and severity of hepatic dysfunction and renal dysfunction

Supplementary note: Hepatic/renal dysfunction means events requiring clinical attention and follow-up, rather than temporary abnormalities in laboratory data.

[6] Creatinine clearance



- [7] Whether the patient is on hemodialysis or not
- [8] Presence/absence of ocular disease history/complications
- [9] Disease history
  - · Name of disease or syndrome
  - Whether the disease is a past one or is present now.

Supplementary note: The name of chronic disease (including allergy), disease requiring treatment, disease or disorder requiring or causing surgery, hospitalization or sequelae, and other possibly problematic disease or syndrome will be recorded. The disease or syndrome seen before the start of treatment with the product is counted as "disease history" and the disease or syndrome present at the start of treatment is counted as "complication."

[10] History of previous treatment drugs for the target disease

(Drugs used during the period from 14 days to 1 day before the start of treatment with the product)

- Name of drug (brand name)
- · Route of administration
- · Daily dose
- · Number of doses per day
- Dosing period
- Reasons for discontinuation
- (3) The following information for the period until the day of safety evaluation will be entered.
  - [1] Pregnancy status and date of delivery/planned date of delivery (females only)

## 6.2 Records of treatment with the product

The following information about the product use until the day of safety evaluation will be entered:

- [1] Daily dose
- [2] Number of doses per day
- [3] Dosing regimen (morning/noon/evening/bedtime, before meal/after meal/others)
- [4] Dosing period

In cases receiving hemodialysis, the following information will be also entered:

- [5] Frequency of dialysis
- [6] Duration of each session of dialysis
- [7] Supplemental dose after dialysis

## 6.3 Concomitant therapy

(1) Drug therapy

The following information will be entered about all drugs used by the day of safety evaluation. If any adverse event occurs, information will be also entered about the concomitant drugs used during the period from the first day of treatment to the onset of the adverse event. Medications used for treatment of the adverse event should be also recorded.

- [1] Name of drug (brand name)
- [2] Route of administration
- [3] Daily dose
- [4] Number of doses per day



- [5] Dosing period
- [6] Reasons for the use of drugs

## (2) Non-drug therapy

The following information will be entered about the non-drug therapies used by the day of safety evaluation. If any adverse event occurs, information will be also entered about the non-drug therapies used during the period from the first day of treatment to the onset of the adverse event. The non-drug therapies used for treatment of the adverse event should be also recorded.

- [1] Name of therapy
- [2] Period of use
- [3] Reason for use

## 6.4 Tests (clinical findings/laboratory test)

## (1) Body weight

The following information will be entered. The body weight will be measured before the start of treatment with the product (including the first day of treatment), at Week 4 and Week 13, and by the day of safety evaluation. If the investigator considers that the change in body weight from the pre-treatment level is abnormal, it will be reported as an adverse event.

- [1] Date of evaluation
- [2] Results

## (2) Clinical findings

The following information will be entered about the clinical findings before the start of treatment (including the first day of treatment) and during the period from the start of treatment to the day of safety evaluation. In cases where treatment has been completed or discontinued before Week 13, the data at the time of completion (discontinuation) of treatment will be entered. If the investigator considers that the change in any of the clinical findings from the pre-treatment status is abnormal, it will be reported as an adverse event.

(2)-1 Information before the start of treatment (including the first day of treatment) and during the period from the start of treatment to the day of safety evaluation

[Presence/absence of peripheral edema or edema in general], [Presence/absence of dizziness, somnolence, loss of consciousness, syncope and potential for accidental injury], [Presence/absence of ophthalmological abnormalities], [Presence/absence of suicidal ideation (including suicide attempt and suicide after start of treatment), [Presence/absence of pathologic changes in appetite and activity]

Supplementary note\*: In cases where peripheral edema or edema in general is found, adverse events of the cardiovascular and respiratory systems also need to be checked. If any clinically significant change from the pre-treatment condition is found, it should be entered in detail in the field for adverse events.

(2)-2 Information in cases of completed (discontinued) treatment with the product (information on the day of safety evaluation following 7-day period after the day of discontinuation [including Day 7 of this period])

[Presence/absence of withdrawal symptom/rebound phenomenon]

## (3) Presence/absence of hyperalgesia

Information will be entered about the presence/absence of hyperalgesia before the start of treatment (including the first day of treatment) and at Week 13. In cases where treatment has been completed or discontinued before Week 13, the data at the time of completion



(discontinuation) of treatment will be entered. If the investigator considers that the change in the condition of hyperalgesia from the pre-treatment status is abnormal, it will be reported as an adverse event.

## (4) Laboratory test

The data on the following laboratory parameters tested before the start of treatment with the product (including the first day of treatment) and during the period from the start of treatment to the day of safety evaluation will be entered. If the investigator considers that the change in any of the following parameters from the pre-treatment level is abnormal, it will be reported as an adverse event.

(Serum creatinine, serum amylase, serum total thyroxine [T4], thyroid stimulating hormone [TSH], blood glucose [fasting level], hemoglobin A1c [HbA1c])

- [1] Date of measurement
- [2] Results

#### 6.5 Clinical evaluation

## (1) Patient-rated pain score

Before the start of treatment (including the first day of treatment) and at Week 4 and Week 13, the pain experienced during the past 24 hours will be rated at the time of getting up in the morning on a 11-grade scale, ranging from 0 (no pain) to 10 (the most severe pain possible). In cases where treatment has been completed or discontinued before Week 13, the data at the time of completion (discontinuation) of treatment will be entered.

## (2) Patient-rated sleep disorder score

Before the start of treatment (including the first day of treatment) and at Week 4 and Week 13, the sleep disorder (inability to sleep because of pain) experienced during the past 24 hours will be rated at the time of getting up in the morning on a 11-grade scale, ranging from 0 (no disturbance of sleep) to 10 (totally unable to sleep because of pain)]. In cases where treatment has been completed or discontinued before Week 13, the data at the time of completion (discontinuation) of treatment will be entered.

### (3) Patient's impression (Patient Global Impression of Change [PGIC])

The patient's impression about the condition at Week 13, as compared to the condition before the start of treatment (including the first day of treatment), will be rated on a 7-grade scale, ranging from 1 (markedly improved) to 7 (markedly worsened). In cases where treatment has been completed or discontinued before Week 13, the data at the time of completion (discontinuation) of treatment will be entered.

- 1. Markedly improved
- 2. Improved
- 3. Slightly improved
- 4. Unchanged

- 5. Slightly worsened
- 6. Worsened
- 7. Markedly worsened

## (4) Physician's impression (Clinical Global Impression of Change [CGIC])

The physician's impression about the condition at Week 13, as compared to the condition before the start of treatment (including the first day of treatment), will be rated on a 7-grade scale, ranging from 1 (markedly improved) to 7 (markedly worsened). In cases where treatment has been completed or discontinued before Week 13, the data at the time of completion (discontinuation) of treatment will be entered.

- 1. Markedly improved
- 2. Improved
- . Slightly improved
- . Unchanged

- 5. Slightly worsened
- Worsened
- 7. Markedly worsened



## 6.6 Patient summary

The appropriateness of continuation of treatment with the product will be checked on the day of safety evaluation. In cases where continuation of treatment with the product is not possible, one major reason should be selected from the alternatives given below. If adverse events, abnormalities in laboratory parameters or the death of patient is selected as a major reason, the relevant data should be entered in the "adverse event" field.

- [1] Insufficient clinical efficacy
- [2] Recovery (effective)
- [3] Adverse events
- [4] Abnormalities in laboratory parameters
- [5] Death of patient
- [6] Lost to follow-up
- [7] Others

In cases where no revisit has been made after the start of treatment, it should be entered in the "Confirmation of revisit after the start of treatment" field.

## 6.7 Efficacy evaluation

The efficacy of the product at Week 13 as compared to the condition before the start of treatment (including the first day of treatment) will be evaluated in the following way, and the judgment will be entered. In cases where treatment has been completed or discontinued before Week 13, the data at the time of completion (discontinuation) of treatment will be entered.

- [1] Date of efficacy evaluation
- [2] Clinical efficacy
  - Effective
  - · Ineffective
  - Impossible to judge (enter the reason)

Items of evaluation

The reason for judging "effective" or "ineffective" should be entered (multiple choices allowed).

- Changes in clinical symptoms
- Others

#### 6.8 Adverse events

For evaluation of safety, the incidence of adverse events following the start of treatment with the product will be checked, and the following information will be entered. If any adverse event occurs, the investigator should take appropriate measures and immediately report it to the sponsor. When the causal relationship between the event and the product cannot be ruled out, observe the course of event or its sequela until they disappear or become stabilized at the level acceptable for the investigator and the sponsor.

A detailed investigation will be separately carried out if patients have intrauterine exposure or develop serious adverse reactions, adverse reactions not listed in the package insert and the like and the sponsor deems it necessary.

- [1] Day of safety evaluation (as a rule, day of last visit within 29 days after the start of treatment)
- [2] Presence/absence of adverse events
- [3] Name of adverse event
- [4] Date of onset
- [5] Measures taken



- [6] Seriousness
- [7] Outcome
- [8] Causal relationship to the product

[The following information should be entered if the adverse event is associated with abnormal changes in test data such as laboratory tests.]

- [1] Name of test
- [2] Reference value at the facility
- [3] Unit
- [4] Date of measurement
- [5] Results

Supplementary note: Adverse events mean all events unfavorable for the patient, arising after the start of treatment with the product, regardless of presence/absence of causal relationship to the product (including clinically significant abnormal changes in laboratory parameters). Serious adverse events mean death, life-threatening events, and events possibly causing hospitalization, extension of hospital stay period, permanent or marked disorders/disabilities, congenital anomalies/defects or other medically significant events/disorders.

## 6.9 Major investigation items

The following events should be evaluated as major investigation items in this survey.

- [1] Peripheral edema and edema-related events
  - Information will be collected about the presence/absence of events related to peripheral edema and the course of patients before and after the onset of events. The situations on development of these events will be analyzed by means of factor analysis, including analysis of the site affected, dose of the product, concomitant therapy, background variables, etc. The package insert gives precautions on congestive heart failure in patients presenting symptoms related to edema. In 30 overseas placebo-controlled studies, the incidence of hypertension and dyspnea was higher in the patients developing peripheral edema than in patients free of peripheral edema, although the incidence of the other events did not differ markedly between these two groups. In view of these facts, information on cardiac function and the incidence of adverse events of the respiratory system will be also collected.
- [2] Dizziness, somnolence, loss of consciousness, syncope and potential for accidental injury

Information will be collected about the presence/absence of events related to dizziness, somnolence, loss of consciousness, syncope and potential for accidental injury and the course of patient's condition before and after the onset of events. The situations on development of these events will be analyzed by factor analysis, including analysis of the dose of the product, concomitant therapy, background variables and so on.

[3] Vision-related events

Information will be collected about the presence/absence of events related to the eyes and the course of patient's condition before and after the onset of events. The situations on development of the events will be analyzed by factor analysis, including analysis of the dose of the product, concomitant therapy, background variables and so on.

Patients developing adverse events included in the major investigation items will be



separately investigated in detail if the sponsor deems it necessary.

## 7 Analysis plan

## 7.1 Analysis set

As a rule, safety analysis set will include patients who satisfy the eligibility criteria and have been confirmed to have taken the product at least once. As a rule, efficacy analysis set will include patients who are evaluable for efficacy in accordance with the separately set analysis plan (i.e., patients in whom efficacy was considered to be appropriately evaluated).

## 7.2 Methods of analysis

## 7.2.1 Safety analysis

In the safety analysis set, the status of onset of adverse reactions and incidence of adverse reactions (percentage of patients developing adverse events for which the causal relationship with the product cannot be ruled out) will be set as primary analysis items. The factors affecting the incidence of adverse reactions will be also analyzed, for example, the incidence of adverse events will be summarized for each of the factors including background variable.

## 7.2.2 Efficacy analysis

In the efficacy analysis set, the response rate will be set as a primary analysis item. As needed, explorative analysis of factors affecting the efficacy will be also carried out.

## 7.3 Time of analysis

## 7.3.1 Periodical safety report

Interim analysis will be conducted at intervals of 6 months during the first two years after approval of the product and once a year during the subsequent reexamination period.

## 7.3.2 Submission of application for reexamination

Final analysis will be conducted upon completion of the reexamination period.

### 8 Publication of the results

Pfizer Japan Inc. will publish the results of one of the following surveys. As needed, the company will publish the results of survey at academic society meetings, in journals and so on for the purpose of supplying information for proper use of the product.

- The survey registered in www.clinicaltrials.gov (ClinicalTrials.gov), regardless of the reason for registration
- Other survey judged to have yielded scientifically or medically significant results

The timing for publication of the survey results will be determined based on whether or not the product has been approved in any country at the completion of the survey on the product. The results of the survey on the product already approved in a given country should be published within one year after fixation of the patient's data collected during the last visit.

Only the published papers which can be accessed via the widely accepted and searchable databases on papers will be cited.

#### 9 Contact information

#### 9.1 Contact information for the contents of survey

| Name | Post-Marketing Surveillance Division, Pfizer Japan Inc. |
|---|---|
| Address | Shinjuku Bunka Quint Building, 3-22-7 Yoyogi, Shibuya-ku, Tokyo 151-8589 |



| Fax | +81-3-5309-9186 |
|--------|--------------------------|
| E-mail | Lyrica EDCMED@pfizer.com |

# 9.2 Contact information for the system

| Name | PostMaNet CSD, Fujitsu FIP Corporation |
|---|---|
| Address | 2-20-5 Shimokodanaka, Nakahara-ku, Kawasaki City, Kanagawa Prefecture 211-8520 |
| Business<br>hours | Monday through Friday, 9:00 a.m. to 9:00 p.m. (excluding national holidays) |
| Tel | +81-120-002-593 |

## 10 References

- Attachment 1: Adverse event report
- Reference 1: Hanaoka K et al., Journal of Pain Clinic 30(10):1395-1408, 2009
   [L20091007038]

